CLINICAL TRIAL: NCT04446169
Title: COVID-19 (SARS-CoV-2) in Urine and Semen: Qualitative and Quantitative Analyses and Evaluation of STD, Sexual Function, Fertility and Urinary Function
Brief Title: COVID-19 (SARS-CoV-2) in Urine and Semen
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Simone Morselli, MD, University of Florence
Other Study IDs: 17104_oss/2020
Record Dates: First submitted 2020-06-20; First posted 2020-06-24 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV 2; Sexual Function and Fertility Disorders; Urinary Function Disorders; Urine; Semen
Keywords: SARS-CoV 2; Sexual Function; Fertility; Urine; Semen
MeSH Terms: interventions — Seeds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV 2 Patients: Patients with previous nasopharyngeal swab positive for SARS-CoV-2, subsequently negativeized in two detections
  Interventions: Diagnostic Test: SARS-CoV 2 RNA PCR Urine; Diagnostic Test: SARS-CoV 2 RNA PCR Semen; Diagnostic Test: Semen Qualitative Analysis; Diagnostic Test: IIEF-5 questionnaire; Diagnostic Test: Male Sexual Health Questionnaire (MSHQ); Diagnostic Test: IPSS questionnaire; Diagnostic Test: SECRET questionnaire; Diagnostic Test: Interleukin assessment in semen

INTERVENTIONS:
Diagnostic Test: SARS-CoV 2 RNA PCR Urine — Search for SARS-CoV 2 RNA in urine through PCR
Diagnostic Test: SARS-CoV 2 RNA PCR Semen — Search for SARS-CoV 2 RNA in Semen through PCR
Diagnostic Test: Semen Qualitative Analysis — Search for Semen Alterations in patients with past SARS-CoV 2 infection
Diagnostic Test: IIEF-5 questionnaire — IIEF-5 assessment in patients with past SARS-CoV 2 infection
Diagnostic Test: Male Sexual Health Questionnaire (MSHQ) — Male Sexual Health Questionnaire (MSHQ) assessment in patients with past SARS-CoV 2 infection
Diagnostic Test: IPSS questionnaire — IPSS assessment in patients with past SARS-CoV 2 infection
Diagnostic Test: SECRET questionnaire — SECRET questionnaire assessment in patients with past SARS-CoV 2 infection
Diagnostic Test: Interleukin assessment in semen — Assessment of Interleukin presence and quantitative analysis in semen, to study if a previous inflammation/infection due to SARS-CoV 2 in testis was present

SUMMARY:
This study is part of the current global emergency scenario due to infection with Coronavirus, SARS-CoV-2 as indicated by the international taxonomy. Study aim is to investigate the possibility of the presence of the virus within the seminal fluid and in the urine of infected patients, both during the acute phase and remotely. Current evidences show that Coronaviruses can be present inside the testicle and sperm in other species, such as in feline and avian models.

In human beings, current researches have mixed results regarding the presence of SARSCoV-2 in urine, as several studies with a large sample found no traces of the same with Real-Time Reverse method Transcriptase - Polymerase Chain Reaction or with method of nucleic acid amplification. By contrast, in just over 6% of 58 patients with Real Time Polymerase Chain Reaction method have found the presence of SARS-CoV-2 in the urine, even at a distance from the last negative nasopharyngeal swab.

Given the topicality of the problem, our study has the objective of specifically researching the presence and possible persistence over time of SARS-CoV-2 in seminal fluid and urine.

A saliva sample will also be collected as a control. At the moment there are no studies in literature that tested this possibility. If confirmed, it would lead to find out another potential method of transmission, the sexual one, in asymptomatic patients or apparently no longer infectious with negative buffer. The rationale for our study is the evidence that in other species this type of transmission by coronaviruses is possible and that at present it has not been verified in mankind.

The relevance of the study would be both in the case of a negative result, as the first study in its generally, both in the case of a positive result, due to the possibility of introducing new prevention measures in the long run.

DETAILED DESCRIPTION:
This study is part of the current global emergency scenario due to infection with Coronavirus, SARS-CoV-2 as indicated by the international taxonomy. Study aim is to investigate the possibility of the presence of the virus within the seminal fluid and in the urine of infected patients, both during the acute phase and remotely. Current evidences show that Coronaviruses can be present inside the testicle and sperm in other species, such as in feline and avian models.

In human beings, current researches have mixed results regarding the presence of SARSCoV-2 in urine, as several studies with a large sample found no traces of the same with Real-Time Reverse method Transcriptase - Polymerase Chain Reaction or with method of nucleic acid amplification. By contrast, in just over 6% of 58 patients with Real Time Polymerase Chain Reaction method have found the presence of SARS-CoV-2 in the urine, even at a distance from the last negative nasopharyngeal swab.

Given the topicality of the problem, our study has the objective of specifically researching the presence and possible persistence over time of SARS-CoV-2 in seminal fluid and urine.

A saliva sample will also be collected as a control. At the moment there are no studies in literature that tested this possibility. If confirmed, it would lead to find out another potential method of transmission, the sexual one, in asymptomatic patients or apparently no longer infectious with negative buffer.

According to results obtained, follow up will be tailored to patients (assessment for COVID 19 infections and/or further analysis/folliow-up in case of abnormal findings) The rationale for our study is the evidence that in other species this type of transmission by coronaviruses is possible and that at present it has not been verified in mankind.

The relevance of the study would be both in the case of a negative result, as the first study in its generally, both in the case of a positive result, due to the possibility of introducing new prevention measures in the long run.

ELIGIBILITY:
Inclusion Criteria:

* Male Sex
* Age>18 years
* Will to participate to the study
* Documented past infection for SARS-CoV2 (Nasopharyngeal swab positive for SARS-CoV2 RNA)
* Current negative infection for SARS-CoV2 (Two negative Nasopharyngeal swab for SARS-CoV2 RNA, done following WHO guidelines)

Exclusion Criteria:

* Age more than 80 years old
* Anejaculation
* Patient's will

Ages: 18 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Semen analysis
Study Population: Prospective cohort study on male patients with a documented previous infection for SARS-CoV2, including symptomatic and asymptomatic patients.Patients need to be eligible for the inclusion criteria and to sign the informed consent to be enrolled to the study
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
SARS-CoV 2 presence in semen | Enrollment
  SARS-CoV 2 RNA PCR in semen
SARS-CoV 2 presence in urine | Enrollment
  SARS-CoV 2 RNA PCR in urine
Inflammation in Semen | Enrollment
  Interleukin quantitative analysis in Semen, to assess if past inflammation due to SARS-CoV 2 Infection was present
Semen quantitative and qualitative analysis | Enrollment
  Spermiogram done following WHO guidelines and criteria

SECONDARY OUTCOMES:
Erectile Function | Enrollment
  International Index of Erectile Function (IIEF-5) questionnaire administration. Score range from 0 to 25. Higher scores mean good erectile function
Sexual Habits | Enrollment
  SExual Chronicle REcording Table (SECRET) questionnaire administration Questionnaire helps to assess the sexual habits of individuals
Urinary function | Enrollment
  International Prostate Symptom Score (IPSS) questionnaire administration Score range from 0 to 35. Higher scores mean worst urinary function
Sexual and Ejaculatory Function | Enrollment
  Male Sexual Health Questionnaire Short Form (MSHQ-SF) admnistration Higher scores mean better sexual and ejaculatory function

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gacci, MD, Principal Investigator — Careggi University Hospital; Sergio Serni, Prof, Study Director — University of Florence
Locations (1):
- AOU Careggi, Florence, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No